CLINICAL TRIAL: NCT06616012
Title: Evaluation of Intravascular Monitoring of Partial PRessure of Oxygen for Neonatal IntensiVE Care Patients -3
Acronym: IMPROVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neosense Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPROVE-3
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Catheters, Indwelling; Preterm Birth; Compromised Health
Keywords: neonatal; arterial oxygen tension; oxygen therapy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neosense Umbilical Catheter (Experimental): The Neosense umbilical catheter is used instead of the routinely used umbilical catheter
  Interventions: Device: Neosense umbilical catheter

INTERVENTIONS:
Device: Neosense umbilical catheter — The Neosense umbilical catheter is used instead of a standard umbilical catheter

SUMMARY:
The study is a non-blinded trial with one single intervention in sick newborn infants. The Neosense umbilical catheter will be used instead of the routinely used umbilical catheter on infants where the treating physician has ordered use of an umbilical catheter. The catheter will be connected to the Neosense monitor/measuring unit.

Blood samples for blood gas analysis are collected from the patients according to the clinical routine (every 4th to 6th hour). Oxygen tension data from the Neosense measuring system, from the time points when a blood gas sample was collected, will be recorded. This data will be compared to the oxygen tension value from the blood gas sample collected at the same time point. The blood gas samples will be analysed according to clinical and laboratory routine.

The infants will remain in the study as long as the Neosense measuring system is used

ELIGIBILITY:
Inclusion Criteria:

Sick newborn infants where the clinical routine indicates use of an umbilical catheter. At least one of the criteria below should be fulfilled:

* The infant needs invasive measurement of blood pressure.
* The infant needs repetitive sampling of blood.
* The infant needs prolonged infusion(s) > 2 days.
* The infant needs infusion of vessel irritating and potentially vessel harming solutions.
* The infant is born extremely preterm (before 28+0 weeks gestational age).
* A newborn infant with severe respiratory disorder, requiring oxygen treatment (more than 40% Fraction of inspired oxygen (FiO2)).
* The infant is undergoing therapeutic hypothermia following asphyxia "oxygen deficiency at birth").
* The infant has a severe infection/sepsis.

Also:

• Signed informed consent form by both parents (or guardians), (if the infant has only one parent (or guardian) one informed consent is required).

Exclusion Criteria:

* Gastroschisis
* Omphalocele
* Peritonitis
* Necrotizing enterocolitis
* Omphalitis
* The infant has a severe infection/sepsis
* Expected MRI investigation within the 7 first days after birth
* The infants birth weight is below 750 g
* The infant is born before week 25+0
* Local vascular compromise in lower limbs or buttocks area, or portal venous hypertension

Ages: 0 Years to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical complications with the Neosense catheter. | During study, up to 5 days
  The number of occasions when the Neosense catheter had to be removed and the underlying reason. This includes all anticipated device effects as well as placing the catheter in the wrong vessel, impossible to measure blood pressure, collect blood samples and/or administer fluids.

SECONDARY OUTCOMES:
Measurement performance (continuously) of an intravascular oxygen sensor in the Neosense system | Measurement comparisons done at every blood gas sample, i.e. every 4th - 6th hour during the study (up to 5 days)
  The oxygen tension measured by the Neosense system, compared to the oxygen tension measured by a blood gas analyser.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sindelar, MD, PhD, Associate professor, Principal Investigator — Uppsala University Children's Hospital
Locations (6):
- Sweden (6):
  - Östra/Sahlgrenska University Hospital, Gothenburg, Halland County
  - Skåne University Hospital, Lund/Malmö, Skåne County
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Södersjukhuset, Stockholm, Stockholm County
  - Uppsala University Children's Hospital, Uppsala, Uppland
  - Västmanalands Hospital, Västerås, Västmanland County

IPD SHARING:
Plan to Share IPD: No